CLINICAL TRIAL: NCT02395562
Title: Association of Viral Reactivation and Skin Cancer in Organ Transplant Recipients
Brief Title: Viral Reactivation and Skin Cancer
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: FUP063
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Skin Cancer; Infection Reactivation
MeSH Terms: conditions — Skin Neoplasms; Latent Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OTR and viral reactivation: Organ transplant recipients with and without viral reactivation and skin cancer

SUMMARY:
Several studies show that the incidence of skin cancer parallels the length and depth of immunosuppression. This study will analyze the correlation of viral reactivation and skin cancer in organ transplant recipients.

DETAILED DESCRIPTION:
Squamous Cell Carcinoma of the skin (SCC) affects people in high numbers worldwide. While a yearly increase of over 2 million patients, who develop cancer, is recorded, organ transplant recipients (OTR) have a 60- to 100-fold higher risk of developing skin cancer. In OTRs, skin cancer is the most frequent tumor that appears, whereas 95% are nonmelanoma skin cancer cells: squamous cells or basal cell carcinomas. All OTRs need to be treated lifelong with immunosuppressants in order to prevent the rejection of the transplanted organ. However, this immunosuppressive treatment leads to a decrease of immunity, and therefore, cancer cells are able to proliferate easier.

Several studies show that the incidence of skin cancer parallels the length and depth of immunosuppression. The appearance of CD4 in OTRs with cutaneous carcinomas is significantly lower compared to those without skin lesions. Various findings have shown a positive correlation of the period of exposure to immunosuppressants and the risk of skin cancer. However, little is known about the dose or the type of drug is responsible for skin cancer. The uptake of three immunosuppressive medicaments compared to the uptake of two results in a 3-fold increased risk of developing cancer. The consequence of the immunosuppressive therapy is reversible; patients who stop immunosuppressive treatment often show a decrease in skin cancer. The highest risk for organ rejection is during the first three months after transplantation. Therefore, an increased dose of immunosuppressors is used during this time.

In addition to cancer, a high increase of viral infections and reactivations is seen in OTRs. Over 90% of the population carries herpesviruses. The risk of viral infection and reactivation is much higher in OTRs. While inducing a decrease in immunosurveillance, herpesvirus can spread easier.

Herpesvirus infections due to the eight human herpes viruses (HHV) are more frequent by immunosuppression in OTRs. Once a patient is infected with one of the human herpesvirus types (Herpes simplex viruses 1 and 2, varicella-zoster virus, Epstein-Barr virus, human cytomegalovirus, human herpesvirus 6 and 7, or Kaposi's sarcoma-associated herpesvirus), the virus is able to establish a latent, non-productive infection and maintains the capacity for a life-long reactivation. Due to the decrease of immunity, OTRs are highly susceptible to activate this latent herpesviral infection, which is a critical aspect of the immunosuppressive treatment. The risk of the reactivation of Cytomegalovirus and Epstein-Barr virus in OTRs is much higher compared to the general population.

Taking the above discussed findings together, the investigators hypothesize that viral infections and reactivations correlate positively with skin cancer in OTRs. Furthermore, the investigators think that viral reactivation and infection can be used as a marker for a later incidence of skin cancer. While virus infections and reactivations appear early, OTRs become affected by SCC in the early and in the late period after the transplantation. The investigators thus aim to analyze existing data from the STCS and its nested studies to test these hypotheses: To assess the correlation of viral replication and skin cancer in organ transplant recipients and to assess viral replication as predictor for skin cancer. The investigators are interested in all data available from other studies of the STCS and to divide all organ transplant recipients e.g. for CMV in four groups: no replication, a larger group who show asymptomatic viral replication, some of them with viral syndrome and the ones with proven disease.

ELIGIBILITY:
Inclusion Criteria:

* oral and written consent to inclusion
* recipient of solid organ transplant

Exclusion Criteria:

* withdrawal of inform consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: organ transplant recipients within the STCS.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2008-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The correlation of skin cancer with viral reactivation in organ transplant recipients | 10 years

SECONDARY OUTCOMES:
The association of viral reactivation and infection in the first year and skin cancer in the following years. Can one be used as a marker for the other one? | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Günther Hofbauer, Prof. MD, Principal Investigator — University Hospital Zurich, Dermatology
Locations (1):
- University Hospital Zurich, Dermatology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
shared with Swiss Transplant Cohort Study. Future projects can obtain data after having a project request approved.